CLINICAL TRIAL: NCT04280198
Title: Using Positive Parent-child Interactions as an Alternative Reinforcer to Promote Healthier Eating Among Young Children
Brief Title: The Play With Me Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Stephanie Anzman-Frasca, Associate Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004200
Record Dates: First submitted 2020-02-18; First posted 2020-02-21 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: High Food Reinforcement; Overeating; Obesity, Childhood
Keywords: relative reinforcing value of food; food reinforcement; positive parenting; parenting intervention
MeSH Terms: conditions — Hyperphagia; Pediatric Obesity

STUDY DESIGN:
Masking Description: Membership in the "intervention" vs. "control" group will not be discussed as such, but participants will know whether they receive intervention activities early (intervention group) or after the post-test assessment (control group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Group 1 - Control (No Intervention): Participants will attend three laboratory visits: baseline 1, baseline 2, and post-test. At baseline 2 and post-test, the primary outcome of child RRV of food vs. parent child interaction is measured. Other measures include child height and weight, child self-regulation, and parenting in the context of a parent-child interaction task. Participants in the control group will not be assigned to complete any intervention activities during the 4-week intervention phase (which takes place between baseline 2 and post-test visits); however, they will receive contacts from a member of the lab each week in the form of electronic reminders (i.e. texts) to remind them of their upcoming post-test laboratory appointment and will receive some intervention materials after the post-test assessment.
- Experimental: Group 2 - Intervention (Experimental): Participants will attend the same three laboratory visits as the control group. The intervention group will also participate in a 4-week intervention, which consists of the parent watching brief weekly parenting videos from the online Triple P Parenting Program and completing interactive parent-child activities from activity boxes created by our laboratory (~60 min of interactive activities/week). Participants will use their activity boxes to practice specific parenting skills from the week's parenting video. Throughout the intervention phase, participants will receive regular text messages to remind them of the week's activities and ask several questions about engagement in study activities over the past 24 hours. The intervention group will also complete an exit interview about the intervention following the post-test assessment to provide insights on fidelity and acceptability.
  Interventions: Behavioral: Triple P Parenting Videos; Behavioral: Activity Boxes

INTERVENTIONS:
Behavioral: Triple P Parenting Videos — Four video clips from the online Triple P Parenting program will be used to promote specific positive parenting practices.
  Arms: Experimental: Group 2 - Intervention
Behavioral: Activity Boxes — There will be about 4 planned activities per week within activity boxes provided to families. The activities will be a context in which the positive parenting behaviors can be practiced. Each activity will take about 15 minutes. Families can pick each week whether they'd like their parenting practice to be embedded in reading activities, nature walks/active games, or arts and crafts. Instructions will be included with each activity, including prompts to allow the parent to apply learnings from that week's parenting video and to allow interactions to be child-led.
  Arms: Experimental: Group 2 - Intervention

SUMMARY:
The obesity epidemic continues to be a major public health concern, with 38% of US adults and 17% of children obese. One factor that has been highlighted as a robust predictor of weight outcomes is the relative reinforcing value (RRV) of food, or how rewarding one finds eating compared to alternative activities. An emerging body of literature has built upon the observed relationship between the RRV of food and weight by hypothesizing that the promotion of alternative reinforcers, or rewarding activities that could take the place of eating, offers a novel approach to decreasing excess energy intake and combatting obesity. We aim to integrate distinct bodies of literature and fill a gap in the evidence by testing whether parenting intervention messages delivered and practiced in the context of shared activities can decrease the RRV of food by making parent-child interactions more rewarding. The ultimate goal of this research is to demonstrate that such an intervention can increase children's motivation to interact with their parent instead of eating a favorite food, demonstrating the potential for positive parent-child interactions to become an alternative source of pleasure.

DETAILED DESCRIPTION:
The modern environment is obesity-promoting, with easy access to palatable, energy-dense foods and appealing sedentary activities. Despite this overarching environment, some individuals are able to maintain a normal weight status, suggesting that there are individual differences in susceptibility to obesity-promoting environments. The RRV of food captures individual differences in the motivation to eat by measuring how hard individuals will work for access to food versus other activities, and it has been shown to predict weight outcomes among infants, children, and adults. In a pilot study with infants, Kong, Eiden, Epstein, et al. demonstrated support for this hypothesis as providing infants and parents with access to group music classes increased infants' reinforcing values of music relative to food. Compared to other age groups, less research has been conducted on the RRV of food in preschool children. Filling this gap in the literature is important, as the preschool period is a period of drastic transitions, including extensive learning of food preferences and habits. Studies have also shown that obesity during adolescence is more likely among children who are already overweight by age 5, further highlighting the importance of innovative approaches to childhood obesity prevention prior to school entry.

In the proposed study, we aim to bring together the literature on food reinforcement and the literature on parenting interventions in early childhood by promoting positive, rewarding parent-child interactions as a novel alternative reinforcer to decrease the RRV of food. Positive parenting can be defined as sensitive, responsive parenting, where parents' responses are appropriate for and contingent upon the child's cues and developmental level. This style of parenting early in life has been linked to positive cognitive and socio-emotional outcomes in adolescence and beyond. The focus of the present study is to assess the initial efficacy of the present parenting intervention, as well as its feasibility. This study will pave the way for future testing of this intervention's effects on the RRV of food and other positive developmental and health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Child is 4-5 years old
* Parent/guardian is 18 years of age or older
* Child is not diagnosed with a serious physical or mental health condition that precludes participation
* At least one of the child's parents/guardians are overweight/obese based on self-reported height and weight. This is intended to facilitate recruitment of children at risk for obesity, given the overarching goals of this research.
* Parent and child are English speaking

Exclusion Criteria:

* The child is outside the age range of 4-5 years
* Child is diagnosed with a serious physical or mental health condition that precludes participation
* Parent/guardian <18 years old
* None of the child's parents/legal guardians overweight/obese based on self-reported height and weight
* Parent or child not English speaking

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Child's relative reinforcing value of food versus parent-child interaction | Week 6 (post-test)
  Computer-based RRV task where child can earn portions of snacks and/or time doing an activity of choice with parent
Change in child's relative reinforcing value of food versus parent-child interaction | Week 2 (baseline), Week 6 (post-test)
  Computer-based RRV task where child can earn portions of snacks and/or time doing an activity of choice with parent
Child's maximum schedule reached for food (food reinforcement) | Week 6 (post-test)
  Computer-based RRV task where child can earn portions of snacks and/or time doing an activity of choice with parent
Change in child's maximum schedule reached for food (food reinforcement) | Week 2 (baseline), Week 6 (post-test)
  Computer-based RRV task where child can earn portions of snacks and/or time doing an activity of choice with parent
Child's maximum schedule reached for parent-child interaction | Week 6 (post-test)
  Computer-based RRV task where child can earn portions of snacks and/or time doing an activity of choice with parent
Change in child's maximum schedule reached for parent-child interaction | Week 2 (baseline), Week 6 (post-test)
  Computer-based RRV task where child can earn portions of snacks and/or time doing an activity of choice with parent

SECONDARY OUTCOMES:
Observations of warm and sensitive parenting | Week 6 (post-test)
  Coded from parent-child interaction using Iowa Family Interaction Rating Scales. The score will be a composite of the following scales, following work by Eiden and colleagues: positive reinforcement, encourages independence, sensitive child-centered, positive mood, warmth/support, prosocial, communication, listener response, relationship quality, rater response. We will also examine relationships between the scales to examine whether the composite is appropriate. Range: 1-9, 9=more warmth/sensitive parenting
Observations of child prosocial behavior | Week 6 (post-test)
  Coded from parent-child interaction using Iowa Family Interaction Rating Scales. Scale: child prosocial behavior. Range: 1-9, 9=more prosocial behavior
Parent-reported nurturance in parenting | Week 6 (post-test)
  Comprehensive General Parenting Questionnaire. Range: 1-5, 5=more nurturance
Parent-reported structure in parenting | Week 6 (post-test)
  Comprehensive General Parenting Questionnaire. Range: 1-5, 5=more structure
Parent-reported nurturance in parenting | Week 10 (follow-up)
  Comprehensive General Parenting Questionnaire. Range: 1-5, 5=more nurturance
Parent-reported structure in parenting | Week 10 (follow-up)
  Comprehensive General Parenting Questionnaire. Range: 1-5, 5=more structure
Parent-reported parenting efficacy | Week 6 (post-test)
  Parenting Sense of Competence Questionnaire. Range: 1-6, 6=more efficacy
Parent-reported parenting efficacy | Week 10 (follow-up)
  Parenting Sense of Competence Questionnaire. Range: 1-6, 6=more efficacy
Parent-reported parenting satisfaction | Week 6 (post-test)
  Parenting Sense of Competence Questionnaire. Range: 1-6, 6=more satisfaction
Parent-reported parenting satisfaction | Week 10 (follow-up)
  Parenting Sense of Competence Questionnaire. Range: 1-6, 6=more satisfaction
Child self-regulation | Week 6 (post-test)
  Head Toes Knees Shoulders Task
Child total behavioral difficulties | Week 6 (post-test)
  Strengths and difficulties questionnaire. Range=0-40, 40=more difficulties
Child overall behavioral difficulties | Week 10 (follow-up)
  Strengths and difficulties questionnaire. Range=0-40, 40=more difficulties
Child prosocial behavior | Week 6 (post-test)
  Strengths and difficulties questionnaire. Range=0-10, 10=more prosocial behavior
Child prosocial behavior | Week 10 (follow-up)
  Strengths and difficulties questionnaire. Range=0-10, 10=more prosocial behavior
Child peer relationships problems | Week 6 (post-test)
  Strengths and difficulties questionnaire. Range=0-10, 10=more peer problems
Child peer relationships problems | Week 10 (follow-up)
  Strengths and difficulties questionnaire. Range=0-10, 10=more peer problems

OTHER OUTCOMES:
Intervention compliance | Week 2-5
  Daily text messages (intervention group only)
Intervention acceptability | Week 2-5
  Daily text messages (intervention group only)
Intervention acceptability | Week 6 (post-test)
  Exit interview (intervention group only)
Intervention use and acceptability | Week 10 (follow-up)
  Parent questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Anzman-Frasca, PhD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- State University of New York at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No